CLINICAL TRIAL: NCT02053064
Title: Long-term Follow-up of Patients With Sanfilippo Type A Syndrome Who Have Previously Been Treated in the P1-SAF-301 Clinical Study Evaluating the Tolerability and Safety of the Intracerebral Administration of SAF-301.
Brief Title: Long-term Follow-up of Sanfilippo Type A Patients Treated by Intracerebral SAF-301 Gene Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LYSOGENE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2-SAF-301
Record Dates: First submitted 2014-01-16; First posted 2014-02-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Mucopolysaccharidosis Type III A; Sanfilippo Disease Type A
Keywords: Neurodegenerative diseases; Nervous systems diseases; Genetic diseases, Inborn; Metabolic diseases; Gene therapy; Adeno Associated Virus (AAV)
MeSH Terms: conditions — Mucopolysaccharidosis III; Neurodegenerative Diseases; Genetic Diseases, Inborn; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SAF-301 (Experimental)
  Interventions: Genetic: SAF-301

INTERVENTIONS:
Genetic: SAF-301

SUMMARY:
P2-SAF-301 is an open-label interventional study without administration of investigational product, evaluating the long-term safety and tolerability of intracerebral SAF-301 previously administered to 4 patients with Sanfilippo type A syndrome.

The primary objective is to collect additional safety and tolerability data on intracerebral SAF-301 previously administered to 4 patients with Sanfilippo type A syndrome.

The secondary objective is to further collect data to assess the effects of SAF-301 on neurological and psychological status, and potential biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients having completed the previous phase I/II study (P1-SAF-301),
* Family understanding the follow-up procedures and the informed consent,
* Patient's parents having signed the informed consent form.

Exclusion Criteria:

* Participation in any other clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Checking of adverse events | until 60 months after SAF-301 administration

SECONDARY OUTCOMES:
Information on neurological and cognitive changes based on clinical status, standardized neurocognitive and behavioral assessments | 5 years after the injection of SAF-301
Information on changes in potential biomarkers of the disease | 5 years after the injection of SAF-301
Information to further evaluation of immune response | 5 years after the injection of SAF-301

CONTACTS AND LOCATIONS:
Overall Officials: Kumaran DEIVA, Dr, Principal Investigator — AP-HP Hôpital Bicêtre
Locations (1):
- Hôpitaux Universitaires Paris Sud (Bicêtre), Le Kremlin-Bicêtre, France